CLINICAL TRIAL: NCT06201845
Title: Assessment of Physical Activity Awareness Training in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-7995
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise awareness training (Experimental)
  Interventions: Other: Exercise awareness training
- physical activity awareness training (Active Comparator): physical activity awareness training,
  Interventions: Other: physical activity awareness training

INTERVENTIONS:
Other: Exercise awareness training — Group exercise training will consist of aerobic exercises including warm-up and cool-down exercises accompanied by music, and trunk strengthening training consisting of core exercises.
  Arms: Exercise awareness training
Other: physical activity awareness training — In the physical activity awareness training, the benefits of exercises on systemic, psychological effects and general body health will be explained and they will be informed about different exercise practice.
  Arms: physical activity awareness training

SUMMARY:
According to the World Health Organization, physical activity is defined as any bodily movement produced by skeletal muscles that requires energy expenditure. Positive effects of leading a physically active life and exercise have been shown in many areas ranging from diabetes to cardiovascular diseases, cancer to mortality, pain to autoimmunity .

DETAILED DESCRIPTION:
Despite the many proven benefits of regular aerobic exercise, physical inactivity remains an important public health problem. In young adults, the perception that exercise is not fun and lack of time for exercise have led to a decrease in physical activity participation . However, studies in the literature have reported that after first creating awareness in individuals about the effects of physical activity on health, creating the necessary time for exercises provides sufficient motivation for individuals to start and continue a more active life.

ELIGIBILITY:
Inclusion criteria:

* 18-25 years of age.
* Being cooperative.
* Voluntarily participating in the study
* Obtaining informed consent from them (Annex-1)

Exclusion criteria:

* Serious musculoskeletal disorders (disc herniation, etc. orthopedic or neurological diagnosis)
* Having a serious systemic disease
* Having a serious injury in the last 3 months.
* Having any neurological problem.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
Jump | 10 weeks
  The jump assesses explosive force through a standing long jump. Participants start from a designated point and jump forward without touching the line, measuring the distance in centimeters from the front of the jumping line to the point where the body's last contact occurred. It's crucial not to lift the feet before jumping, and at least two attempts are made to achieve the best distance.
Grip Strength Assessment | 10 weeks
  Using a JAMAR hand dynamometer, grip strength for both dominant and non-dominant hands is measured during isometric contractions. Participants sit with shoulder adduction, elbow at 90° flexion, and forearm and wrist in a neutral position, gripping and squeezing the dynamometer with maximum force. The test is repeated three times, recording the highest reading in kilograms of force.
Plank Test | 10 weeks
  Assesses the control, strength, and endurance of stabilizing core and back muscles. It's a vital exercise for training the endurance of rectus abdominis and external oblique abdominis muscles. The test shows excellent reliability in evaluating core strength and endurance
Modified Closed Kinetic Chain Upper Extremity Stability Test | 10 weeks
  This test identifies deficits in functional performance of the upper extremity in closed kinetic chain positions. It involves a person assuming a push-up position and rapidly touching one hand's dorsal side to the other hand's dorsum within 15 seconds, aiming to maintain parallel alignment with the ground. The evaluator counts the correct hand touches, and the average of three maximal attempts determines the score.

SECONDARY OUTCOMES:
Sit-Up Test | 10 weeks
  Measures abdominal muscle endurance by performing as many sit-ups as possible within 60 seconds. Participants lie on their backs, knees slightly bent, and hands placed parallel to the ground with palms facing downwards. They aim to touch their knees with their elbows while lifting their upper body without support from the hands

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçehir University, Istanbul, Turkey (Türkiye)